CLINICAL TRIAL: NCT00776906
Title: Advance® 18PTX® Balloon Catheter Study: Treatment of Lesions in Superficial Femoral Artery/Popliteal Artery With a Paclitaxel-coated Balloon
Brief Title: Advance® 18PTX® Balloon Catheter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-008; 190007, PCBS
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2014-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (2):
- 1 (Experimental): PTX-coated balloon
  Interventions: Device: Advance® 18PTX® Balloon Catheter
- 2 (Active Comparator): Bare balloon
  Interventions: Device: Advance® 18LP Balloon Catheter

INTERVENTIONS:
Device: Advance® 18PTX® Balloon Catheter
  Arms: 1
Device: Advance® 18LP Balloon Catheter
  Arms: 2

SUMMARY:
The Advance® 18 PTX® Balloon Catheter study is a clinical trial to study the safety and effectiveness of the Advance 18® PTX® Balloon Catheter in the treatment of lesions in the superficial femoral artery and popliteal artery.

ELIGIBILITY:
Key Inclusion Criteria:

* Age >18 years.
* Able to provide informed consent.
* Has at least one de novo or restenotic lesion(s) with > 70% stenosis documented angiographically of the SFA or popliteal artery. If more than one lesion requires intervention, only one should be treated as a study lesion.

Key Exclusion Criteria:

* Has significant stenosis (> 50%) or occlusion of inflow tract (proximal ipsilateral, iliofemoral, or aortic lesions) not successfully treated before this procedure.
* Lack of at least one patent runoff vessel with < 50% stenosis throughout its course.
* Lesions in target area requiring atherectomy (or ablative devices), cutting balloons, cryoplasty balloons, or any other advanced device to facilitate angioplasty balloon or stent delivery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of Late Lumen Loss | 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (3):
  - Heart Center Leipzig/Park Hospital, Leipzig
  - Klinikum Rosenheim, Rosenheim
  - Universitat Klinik Tubingen, Tübingen
- Endosurgery and Lithotripsy Center, Moscow, Russia